CLINICAL TRIAL: NCT03616418
Title: Ankle Brachial Index Combined With Serum Uric Acid Levels Improve Prediction All Cause Mortality and Cardiovascular Mortality in the Elderly Chinese Population
Acronym: abilities
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, cardiology department of shanghai 10th people's hospital, Shanghai 10th People's Hospital
Other Study IDs: abilities
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Ankle Brachial Index
Keywords: ankle brachial index; cardiovascular disease; risk factors; Framingham Cardiovascular Risk Score; uric acid; survival analysis
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: antiplatelet drugs;statins;antihypertensive drugs
  Other Names: According to the international guidelines, we treated patients who suffered from different disease.

SUMMARY:
Peripheral arterial disease (PAD) is a common clinical manifestation of the systemic atherosclerotic process, and the ankle brachial index (ABI) is an ideal tool to diagnose PAD. The association between high serum uric acid levels (SUA) and arterial stiffness as well as endothelial dysfunction has been demonstrated in humans and uric acid has been suggested to be an important modulator of the inflammatory process. It has also been confirmed by clinical studies. Currently, there have been few long term follow up studies focused on the whether serum uric acid levels combined with ankle brachial index can improve prediction all cause mortality and cardiovascular mortality,especially in China population.Therefore, the aim of this study was to elucidate whether ABIcombined with SUA can improve prediction all cause mortality and cardiovascular mortality in the elderly China population independently of the traditional Framingham Risk Score.

DETAILED DESCRIPTION:
This study is a prospective community-based cohort study, which is aimed to investigate the prognostic factors, including conventional cardiovascular risk factors and measure ABI,SUA,asymptomatic target organ damage, for mortality and cardiovascular diseases. All population were separated into ABI ≤0.50，0.51 <ABI ≤0.9，and 0.91 <ABI≤1.40 three groups according to the ABI. ABI ≤0.9 was selected as cut point for the definition of PAD. Factors related to CVD and all-cause mortality, major adverse cardiac events (MACE) during follow-up was observed by multivariate Cox regression analysis and log rank test. Potential confounding variables with P <0.10 were adjusted for multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

1. age≥65 years old
2. Shanghai residents
3. Sign informed consent

Exclusion Criteria:

1. serious heart disease (NYHA>IV) or end stage renal disease (CKD > 4)
2. cancer and life expectancy was less than 5 years
3. Severe congestive heart failure and Severe renal failure patients
4. Participants had other diseases that required withdrawal from the clinical trial
5. Patients are reluctant to participate in clinical research
6. The patient violated the experimental protocol
7. Clinical diagnosis of Alzheimer's Disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: subjects aged over 65 years old, living in communities located in the Shanghai, will be invited to participate in the present study, if they are willing to give their written informed consents.
Sampling Method: Probability Sample
Enrollment: 3026 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
all cause mortality and cardiovascular mortality | From August 2018 to August 2020
  Cardiovascular events definitions: Hospitalized myocardial infarction was classified as definite or probable based on chest pain symptoms, cardiac enzyme levels, and electrocardiographic findings, or angioplasty28. Coronary heart disease was determined to be present if there was (1) electrocardiographic (ECG) evidence of a prior myocardial infarction, (2) prior coronary artery bypass surgery or angioplasty, (3) Coronary angiography show coronary heart disease, (4) have symptoms of angina and ECG revealed myocardial ischemia performance or laboratory tests showed cardiac enzymes increased and exclude other types of disease, (5) a self-reported history of a physician-diagnosed heart attack 29. CHD death was classified "definite" based on chest pain symptoms, hospital records, and medical history.

IPD SHARING:
Plan to Share IPD: No